CLINICAL TRIAL: NCT03921502
Title: Randomized Multicentre Double-blind Clinical Trial Comparing ERCP vs ERCP and Transmural Gall Bladder Drainage in Non-surgical Patients With Symptomatic Choledocholithiasis
Brief Title: Clinical Trial Comparing ERCP vs ERCP and Transmural Gall Bladder Drainage
Acronym: PECAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Marina de Benito Sanz, Principal investigator, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2019-04-13; First posted 2019-04-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Bile Duct; Obstruction, With Calculus; Choledocholithiasis
Keywords: Choledocholithiasis; Gall Bladder drainage; LAMS
MeSH Terms: conditions — Bites and Stings; Choledocholithiasis | interventions — laminin beta2

STUDY DESIGN:
Intervention Model Description: Multicentric double-blind randomized trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient and the physician responsible for the follow-up will be blinded as to the procedure performed (it will not be specified if transmural drainage was performed in the endoscopic report, nor will images of the drainage be included in the discharge report available in the electronic medical record until after the completion of the study or if complications are suspected).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCP with sphincterotomy + gall bladder drainage with LAMS (Experimental): An ERCP with biliary sphincterotomy will be performed. The performance of other techniques (balloon extraction, dilation, placement of biliary prosthesis ...) is at the expense of the endoscopist. After this, transmural drainage of the gallbladder will be performed by placing a LAMS Axios (Boston Scientific) usually 15x10 mm or 10x10 mm to allow direct cholecystoscopy with a conventional gastroscope or transnasal gastroscope. The placement of the drainage will be performed in the same endoscopic act, by means of an Olympus® sectorial echoendoscope, assisted with X-rays, which allows puncturing the vesicle from the gastric antrum or the duodenal bulb to generate a cholecysto-gastrostomy or cholecysto-duodenostomy respectively. After the puncture of the vesicle from the most optimal anatomical point, it will be tutored with guidance and a Hot Axios® PAL will be placed on it to generate the anastomosis between the aforementioned structures.
  Interventions: Procedure: Gall bladder transmural drainage with LAMS
- ERCP with sphincterotomy (Active Comparator): An ERCP with biliary sphincterotomy will be performed. The performance of other techniques (balloon extraction, dilation, placement of biliary prosthesis ...) is at the expense of the endoscopist.
  Interventions: Procedure: Gall bladder transmural drainage with LAMS

INTERVENTIONS:
Procedure: Gall bladder transmural drainage with LAMS — Placing a PAL Axios (Boston Scientific) usually 15x10 mm or 10x10 mm to allow direct cholecystoscopy with a conventional gastroscope or transnasal gastroscope. The placement of the drainage will be performed in the same endoscopic act, by means of an Olympus® sectorial echoendoscope, assisted with X-rays, which allows puncturing the vesicle from the gastric antrum or the duodenal bulb to generate a cholecysto-gastrostomy or cholecysto-duodenostomy respectively. After the puncture of the vesicle from the most optimal anatomical point, it will be tutored with guidance and a Hot Axios® PAL 15x10 mm or 10x10 mm will be *placed on it to generate the anastomosis between the aforementioned structures.

SUMMARY:
Cholelithiasis occurs in 10-20% of the general population. Up to 18% of these subjects will present symptoms. In patients with symptomatic choledocholithiasis who are not candidates for surgery with indication for ERCP, transmural drainage of the gallbladder reduces the risk of recurrence.

The investigators propose a multicentric double-blind randomized trial. Our primary objective is to assess whether ERCP associated with transmural gallbladder drainage is able to reduce biliary disease income compared with ERCP in patients not candidates for surgery with symptomatic choledocholithiasis and cholelithiasis during one year of follow-up. Also the investigators will analyze the proportion of technical success and complications.

The study population includes all patients older than 75 years with symptomatic choledocholithiasis. An estimated 75 subjects per group (ERCP alone and ERCP and transmural drainage) are needed.

DETAILED DESCRIPTION:
1. Introduction Cholelithiasis occurs in 10-20% of the general population (1). Up to 18% of these subjects will present symptoms and, of these, 1.5% will present an episode of pancreatitis, cholecystitis or acute cholangitis (2). In this way, the pathology associated with biliary lithiasis is the first digestive cause of hospital admission (3).

   The treatment of the pathology associated with biliary lithiasis therefore deals with two problems, controlling the acute process and preventing new episodes. In general, laparoscopic cholecystectomy is the recommended method to reduce the risk of recurrence.
2. Hypothesis

   Conceptual hypothesis:

   In patients with symptomatic choledocholithiasis who are not candidates for surgery with indication for ERCP, transmural drainage of the gallbladder reduces the risk of recurrence.

   Operational hypothesis:

   In subjects> 75 years with symptomatic choledocholithiasis, performing an ERCP with sphincterotomy and transmural drainage of the gallbladder vs. ERCP with sphincterotomy reduces the risk of admission due to complications of cholelithiasis during a 1-year follow-up period.
3. Objectives.

   Primary objective:

   - To assess whether ERCP associated with transmural gallbladder drainage is able to reduce biliary disease income compared with ERCP in patients not candidates for surgery with symptomatic choledocholithiasis and cholelithiasis during one year of follow-up.

   Secondary objectives:
   * Describe the proportion of technical successes and complications associated with transmural biliary drainage, ERCP and those associated with admission.
   * Compare the proportion of income from non-biliary causes in both groups.
   * Compare mortality during admission and during follow-up in both groups.
   * To compare the incidence of biliary and non-biliary admissions during the follow-up year in both groups.
   * Compare the hospital costs of the index income and those generated in the 12 months of follow-up between the patients assigned to the control group and the experimental group.
4. Design Multicentric double-blind randomized trial
5. Methods Study population The study population includes all patients older than 75 years with symptomatic choledocholithiasis. This includes the pictures of acute cholangitis, obstructive jaundice or biliary colic secondary to choledocholithiasis. Participation in the study will be offered to all consecutive patients who meet inclusion criteria and do not present exclusion criteria diagnosed in the participating centers once the project is started until the estimated sample size is completed (see below). Given that in these patients the usual clinical practice is the realization of an ERCP, they will be identified from the ERCP requests received in the endoscopy units.

Intervention Patients who meet the inclusion criteria and do not present any exclusion criteria will be invited to participate in the study. Between the formalization of the request and the endoscopic exploration the informed consent will be completed according to the law 41/2002 of autonomy of the patient without that for that reason the relationship with his doctor is altered or there is any prejudice in his treatment.

1. Endoscopic act

   It will be held at the Rio Hortega University Hospital, the University General Hospital of Alicante or the Ramón y Cajal University Hospital. First, ERCP will be performed. Subsequently, an endoscopic ultrasound will be performed to rule out local causes of exclusion. If there is no contraindication, randomization and placement of transmural vesicular drainage will be carried out if assigned to the intervention group:
   * Control group: An ERCP with biliary sphincterotomy will be performed. The performance of other techniques (balloon extraction, dilation, placement of biliary prosthesis ...) is at the expense of the endoscopist. The procedure will be performed under direct sedation with propofol controlled by the endoscopist team, and with CO2 (carbon dioxide) insufflation.
   * Intervention group: ERCP with biliary sphincterotomy will be performed. The performance of other techniques (balloon extraction, dilation, placement of biliary prosthesis ...) is at the expense of the endoscopist. After this, transmural drainage of the gallbladder will be performed by placing a LAMS (lumen apposing metal stent) Axios (Boston Scientific) usually 15x10 mm or 10x10 mm to allow direct cholecystoscopy with a conventional gastroscope or transnasal gastroscope. The placement of the drainage will be performed in the same endoscopic act, by means of an Olympus® sectorial echoendoscope, assisted with X-rays, which allows puncturing the vesicle from the gastric antrum or the duodenal bulb to generate a cholecysto-gastrostomy or cholecysto-duodenostomy respectively. After the puncture of the vesicle from the most optimal anatomical point, it will be tutored with guidance and a Hot Axios® LAMS will be placed on it to generate the anastomosis between the aforementioned structures. After the placement of the prosthesis, it will be subject to the decision of the endoscopist to perform cholescystoscopy to perform the maneuvers it deems appropriate (extraction of stones, taking biopsies, resection of polyps ...). The performance of both procedures will be performed under direct sedation with propofol controlled by the endoscopist team, and with CO2 insufflation, according to the usual practice of the HURH (Universitary Hospital Río Hortega) Endoscopy Unit.
2. Hospitalization:

After the procedure, the hospital management is in the hands of its responsible physicians in plant at the requesting center. A report will be delivered that does not show if the patient has had the LAMS implanted or not. Therefore, physicians responsible for plant management will not receive information about the assigned group or whether transmural vesicular drainage has been performed.

C.3) Follow-up:

It will be held in each of the participating centers. It will consist of 4 face-to-face visits (after 1 day, 3 months, 6 months and 12 months after the procedure) and 2 phone calls (7 days after the procedure and 9 months). In the case of institutionalized patients or those with serious mobility problems, in-person visits may be made by telephone in an exceptional manner. The physician responsible for the follow-up will be blinded as to the procedure performed (it will not be specified if transmural drainage was performed in the endoscopic report, nor will images of the drainage be included in the discharge report available in the electronic medical record until after the completion of the study or if complications are suspected). During the follow-up visits, it will be confirmed that the prosthesis remains normalized by abdominal ultrasound.

Sample size Assuming a proportion of readmissions of biliary cause of 25% in the control group and 7% in the experimental group, with an alpha risk of 5% and a power of 80% and using the arc transformation sine given the proportion of the experimental group, an estimated 60 subjects per group are needed. Given the age of the patients to be included and the mortality associated with the underlying disease, a proportion of losses of 20% is estimated, which would require 75 patients per group. The annual number of ERCP performed at the Río Hortega university hospital ranges from 1,000 to 1100. Assuming also a number of examinations to be carried out in the collaborating centers, with the inclusion and exclusion criteria exposed, a recruitment interval of 12-18 months is estimated.

Randomization It will be done once the patient agrees to participate in the work and has verified the absence of exclusion criteria. To avoid imbalances between the groups, it will be stratified by baseline diagnosis (cholangitis vs others), given that the mortality during admission associated with acute cholangitis is significantly greater than in the rest of the included conditions. Within each stratum a pure randomization will be carried out by means of a sequence generated by computer where the probability of belonging to each group will be 0.5. For each stratum, there will be a total of n numbered closed opaque envelopes (where n = total sample size) that will be stored in the endoscopy unit and will be opened consecutively as participants are included.

Adverse effects monitoring The adverse effects identified during the study will be classified according to the classification of ASGE (for adverse endoscopic effects) for those associated with hospitalization. According to the interval from the procedure they will be divided between postprocedure (in the first 7 days from the same) and late (after this time). Its relationship with the procedure will be classified as definitive, probable, possible or improbable.

Data Collect The data collection will be done by the main researcher or collaborating researchers through a data collection notebook (CRD) anonymously and dissociated from the clinical information by means of a patient identification code.

6. Data management Data from the data collection notebooks will be merged by the main researcher or collaborating researchers anonymously, encrypted and decoupled from the clinical information by means of a patient identification code (ID), in a database made through the application RedCap available through the Spanish Association of Gastroenterology and the data will be downloaded in the form of an Excel file (Microsoft Corporation,USA). The responsible researcher will define an ID for each participant. The data entered in the database will be anonymous and the database will be protected with a password to which only the researchers will have access.

The unified file will be kept in the Río Hortega University Hospital and will be maintained until the end of the study. Regarding the application of the Organic Law on Data Protection 15/1999 and Royal Decree 1720/2007 that develops it, it should be noted that the protocol defined in the project oriented to epidemiological analysis, determines that the files will record information completely anonymized.

7. Statistical analysis It will be done through the STATA program (StataCorp, 2013. Stata Statistical Software: Release 13. College Station, StataCorp LP).

Descriptive analysis In the quantitative variables the arithmetic average and the standard deviation will be calculated (the variables that do not follow a normal distribution will be described with median, minimum, maximum and interquartile range), and the categorical ones will be expressed as percentages and their 95% confidence intervals .

Hypothesis contrast The analysis of the primary objective, the hospital admission of biliary cause, will be carried out through the Z test of homogeneity without using the correction of Yates. The confidence interval of the difference between the two groups will also be estimated. An intention-to-treat analysis will be performed, regardless of the endoscopic treatment received after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic choledocholithiasis (choledocholithiasis demonstrated radiologically or highly suspected by clinical data (acute cholangitis or obstructive jaundice), analytical and imaging according to the criteria of high probability of choledocholithiasis established in the clinical guidelines (ASGE Guide).
* Discarded for surgical treatment due to age, comorbidity or refusal of the patient.
* Age>75 years

Exclusion Criteria:

* Charlson comorbidity scale adjusted to age <4.
* Hepatobiliary surgery or previous superior digestive tract.
* Ascitis.
* Inability to tolerate sedation of endoscopy, perforation of the digestive tract or other contraindication to endoscopy.
* Coagulopathy with INR (international normalized ratio) > 1.5 not correctable or thrombocytopenia <50000 / mm3 not correctable.
* Other diagnoses at admission (acute cholecystitis, acute pancreatitis, biliopancreatic neoplasia).
* Hemodynamic instability.
* Urgent procedure performed after hours
* No availability of expert material / endoscopist in drainage.
* Anatomical impossibility of performing biliary drainage (absence of vesicular distension, contact between gallbladder and stomach or duodenum, contact area <10 mm).
* Baseline ECOG (Easthern Cooperative Oncology Group) > = 4
* Expectancy of survival <6 months.
* Refusal to participate.
* Distance between the gallbladder and upper digestive tract> 1cm, scleroatrophic vesicle, lack of stable acoustic window for drainage
* ERCP failed (inhability to dain common bile duct)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of paticipants readmitted due to biliary pathology | 1 year
  Rate of participants readmitted due to biliary pathology (cholecystitis, cholangitis, pancreatitis, hepatic abscess...) in each group

SECONDARY OUTCOMES:
Number of participants with technical success | 1 day
  Number of participants with correct placement of the stent from the gastric or duodenal lumen to the gallbladder, together with the documentation of bile flow and / or contrast through it.
Number of dead participants | 1 year
  Rate of deaths in each group
Hospital costs (euros) | 1 year
  Hospital costs (euros) during the period of follow up, including the baseline admission

CONTACTS AND LOCATIONS:
Overall Officials: Ana Y Carbajo López, MD, Principal Investigator — Hospital Río Hortega
Locations (1):
- Hospital Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee TH, Park DH, Lee SS, Seo DW, Park SH, Lee SK, Kim MH, Kim SJ. Outcomes of endoscopic transpapillary gallbladder stenting for symptomatic gallbladder diseases: a multicenter prospective follow-up study. Endoscopy. 2011 Aug;43(8):702-8. doi: 10.1055/s-0030-1256226. Epub 2011 Mar 21. PMID 21425042
- [Background] Choi JH, Lee SS, Choi JH, Park DH, Seo DW, Lee SK, Kim MH. Long-term outcomes after endoscopic ultrasonography-guided gallbladder drainage for acute cholecystitis. Endoscopy. 2014 Aug;46(8):656-61. doi: 10.1055/s-0034-1365720. Epub 2014 Jun 30. PMID 24977397
- [Background] Walter D, Teoh AY, Itoi T, Perez-Miranda M, Larghi A, Sanchez-Yague A, Siersema PD, Vleggaar FP. EUS-guided gall bladder drainage with a lumen-apposing metal stent: a prospective long-term evaluation. Gut. 2016 Jan;65(1):6-8. doi: 10.1136/gutjnl-2015-309925. Epub 2015 Jun 3. No abstract available. PMID 26041748
- [Background] Kahaleh M, Perez-Miranda M, Artifon EL, Sharaiha RZ, Kedia P, Penas I, De la Serna C, Kumta NA, Marson F, Gaidhane M, Boumitri C, Parra V, Rondon Clavo CM, Giovannini M. International collaborative study on EUS-guided gallbladder drainage: Are we ready for prime time? Dig Liver Dis. 2016 Sep;48(9):1054-7. doi: 10.1016/j.dld.2016.05.021. Epub 2016 Jun 3. PMID 27328985
- [Background] de la Serna-Higuera C, Perez-Miranda M, Gil-Simon P, Ruiz-Zorrilla R, Diez-Redondo P, Alcaide N, Sancho-del Val L, Nunez-Rodriguez H. EUS-guided transenteric gallbladder drainage with a new fistula-forming, lumen-apposing metal stent. Gastrointest Endosc. 2013 Feb;77(2):303-8. doi: 10.1016/j.gie.2012.09.021. Epub 2012 Dec 1. No abstract available. PMID 23206813
- [Background] McCarthy ST, Tujios S, Fontana RJ, Rahnama-Moghadam S, Elmunzer BJ, Kwon RS, Wamsteker EJ, Anderson MA, Scheiman JM, Elta GH, Piraka CR. Endoscopic Transpapillary Gallbladder Stent Placement Is Safe and Effective in High-Risk Patients Without Cirrhosis. Dig Dis Sci. 2015 Aug;60(8):2516-22. doi: 10.1007/s10620-014-3371-4. Epub 2014 Oct 7. PMID 25287001
- [Background] Itoi T, Sofuni A, Itokawa F, Tsuchiya T, Kurihara T, Ishii K, Tsuji S, Ikeuchi N, Tsukamoto S, Takeuchi M, Kawai T, Moriyasu F. Endoscopic transpapillary gallbladder drainage in patients with acute cholecystitis in whom percutaneous transhepatic approach is contraindicated or anatomically impossible (with video). Gastrointest Endosc. 2008 Sep;68(3):455-60. doi: 10.1016/j.gie.2008.02.052. Epub 2008 Jun 17. PMID 18561927
- [Background] Sodergren MH, Markar S, Pucher PH, Badran IA, Jiao LR, Darzi A. Safety of transvaginal hybrid NOTES cholecystectomy: a systematic review and meta-analysis. Surg Endosc. 2015 Aug;29(8):2077-90. doi: 10.1007/s00464-014-3915-x. Epub 2014 Nov 26. PMID 25424364
- [Background] McGillicuddy EA, Schuster KM, Barre K, Suarez L, Hall MR, Kaml GJ, Davis KA, Longo WE. Non-operative management of acute cholecystitis in the elderly. Br J Surg. 2012 Sep;99(9):1254-61. doi: 10.1002/bjs.8836. Epub 2012 Jul 24. PMID 22829411
- [Background] Garcia-Alonso FJ, de Lucas Gallego M, Bonillo Cambrodon D, Algaba A, de la Poza G, Martin-Mateos RM, Bermejo F. Gallstone-related disease in the elderly: is there room for improvement? Dig Dis Sci. 2015 Jun;60(6):1770-7. doi: 10.1007/s10620-014-3497-4. Epub 2015 Jan 11. PMID 25577265
- [Background] Trust MD, Sheffield KM, Boyd CA, Benarroch-Gampel J, Zhang D, Townsend CM Jr, Riall TS. Gallstone pancreatitis in older patients: Are we operating enough? Surgery. 2011 Sep;150(3):515-25. doi: 10.1016/j.surg.2011.07.072. PMID 21878238
- [Background] Prevalence of gallstone disease in an Italian adult female population. Rome Group for the Epidemiology and Prevention of Cholelithiasis (GREPCO). Am J Epidemiol. 1984 May;119(5):796-805. PMID 6720676
- [Background] Itoi T, Tsuyuguchi T, Takada T, Strasberg SM, Pitt HA, Kim MH, Belli G, Mayumi T, Yoshida M, Miura F, Buchler MW, Gouma DJ, Garden OJ, Jagannath P, Gomi H, Kimura Y, Higuchi R; Tokyo Guideline Revision Committee. TG13 indications and techniques for biliary drainage in acute cholangitis (with videos). J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):71-80. doi: 10.1007/s00534-012-0569-8. PMID 23307008
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Riall TS, Zhang D, Townsend CM Jr, Kuo YF, Goodwin JS. Failure to perform cholecystectomy for acute cholecystitis in elderly patients is associated with increased morbidity, mortality, and cost. J Am Coll Surg. 2010 May;210(5):668-77, 677-9. doi: 10.1016/j.jamcollsurg.2009.12.031. PMID 20421027
- [Background] Peery AF, Crockett SD, Barritt AS, Dellon ES, Eluri S, Gangarosa LM, Jensen ET, Lund JL, Pasricha S, Runge T, Schmidt M, Shaheen NJ, Sandler RS. Burden of Gastrointestinal, Liver, and Pancreatic Diseases in the United States. Gastroenterology. 2015 Dec;149(7):1731-1741.e3. doi: 10.1053/j.gastro.2015.08.045. Epub 2015 Aug 29. PMID 26327134
- [Background] McSherry CK, Ferstenberg H, Calhoun WF, Lahman E, Virshup M. The natural history of diagnosed gallstone disease in symptomatic and asymptomatic patients. Ann Surg. 1985 Jul;202(1):59-63. doi: 10.1097/00000658-198507000-00009. PMID 4015212
- [Background] Kratzer W, Mason RA, Kachele V. Prevalence of gallstones in sonographic surveys worldwide. J Clin Ultrasound. 1999 Jan;27(1):1-7. doi: 10.1002/(sici)1097-0096(199901)27:13.0.co;2-h. PMID 9888092

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT03921502/Prot_SAP_000.pdf